CLINICAL TRIAL: NCT06793709
Title: Post-marketing Observational Study of Tasfygo Tablet 35 mg to Evaluate the Safety of Tasfygo in Patients With Unresectable Biliary Tract Cancer With FGFR2 Fusion Gene Positivity Who Progressed After Chemotherapy
Brief Title: A Post-marketing Observational Study of Tasfygo in Participants With Unresectable Biliary Tract Cancer With Fibroblast Growth Factor Receptor 2 (FGFR2) Fusion Gene Positivity Who Progressed After Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7090-M081-501
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-01

CONDITIONS: Biliary Tract Cancer
Keywords: Tasfygo; FGFR2 fusion; Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tasfygo tablet 35 milligrams (mg)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary purpose of this study is to investigate the safety of Tasfygo.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with unresectable biliary tract cancer with FGFR2 fusion gene positivity who are naïve to Tasfygo tablet and progressed after chemotherapy.

Exclusion Criteria:

Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with FGFR2 fusion positive unresectable biliary tract cancer with prior chemotherapy who will receive Tasfygo tablet as per daily practice and package insert will be enrolled.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2030-11-12 (Estimated); Study Completion 2030-11-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Drug Reactions | Up to 1 year

SECONDARY OUTCOMES:
Percentage of Participants With Best Overall Response (BOR) Based on Physician's Assessment | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- #Eisai Trial Site 1, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.